CLINICAL TRIAL: NCT03849534
Title: Evaluation of Different Treatment Modalities in Children With Myalgia or Arthralgia in the Temporomandibular Region - a Randomized, Single-blinded, Controlled Non-inferiority Study
Brief Title: Treatment of Temporomandibular Disorders in Children and Adolsecents
Acronym: TMD/PED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Folktandvården Stockholms län AB (Other Government)
Responsible Party: Principal Investigator, Nikolaos Christidis, Associate professor, Senior Lecturer, Senior Consultant, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BettfysPed
Record Dates: First submitted 2019-02-20; First posted 2019-02-21 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Temporomandibular Disorder; Myalgia; Arthralgia of TMJ
Keywords: Children; Mixed dentition; Primary dentition; Adolescents; Myalgia; Arthralgia of TMJ; Treatment; Side-effects
MeSH Terms: conditions — Temporomandibular Joint Disorders; Myalgia | interventions — Counseling

STUDY DESIGN:
Intervention Model Description: Non-inferiority study with two patient arms that are randomized to one of three different treatment arms.
  75 children with TMD myalgia are randomized to one of three treatment arms 75 children with TMD arthralgia are randomized to one of three treatment arms
Who Masked: Investigator
Masking Description: The investigator is blinded to treatment that is performed by a specialist in orofacial pain. The patient is instructed to not reveal the treatment to the investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Soft occlusal appliance (Active Comparator): Individually casted appliances
  Interventions: Device: Soft occlusal appliance; Behavioral: Jaw exercises; Behavioral: Counseling
- Jaw exercises (Active Comparator): Resistance exercises to do twice a day
  Interventions: Device: Soft occlusal appliance; Behavioral: Jaw exercises; Behavioral: Counseling
- Counseling (Active Comparator): Just information at the first visit
  Interventions: Device: Soft occlusal appliance; Behavioral: Jaw exercises; Behavioral: Counseling

INTERVENTIONS:
Device: Soft occlusal appliance — According to Best Practice in Sweden the soft occlusal appliance is ranked as gold standard for children with mixed or primary dentition
Behavioral: Jaw exercises — The participants do three exercises twice a day. Open and closing mouth against resistance as well as stretch
Behavioral: Counseling — The patients are instructed to minimize jaw parafunctions, chewing chewing gum etc, to do exercises, to take pain-killers or NSAIDs etc.

SUMMARY:
Children and adolescents are treated with routine treatment approaches for adults and one of the most commonly used treatments are occlusal appliances. The use of occlusal appliances in managing orofacial pain conditions is supported by evidence, but only for adults. However, the efficacy of the treatment approaches and any possible side-effects/impairment of mandibular growth are absent.

Therefore, the aim of this project is to investigate the effectiveness and possible side-effects of different treatment modalities, such as an occlusal appliance, jaw exercises, NSAID for the conditions myalgia orarthralgia in the orofacial region in children with primary or mixed dentition.

DETAILED DESCRIPTION:
It is well known that the impact of pain in the orofacial region is not only the unpleasant sensory experience but also an emotional experience with feelings of failure, misery, guilt, alienation, and co-morbid depression. TMD is a collective term embracing chronic pain conditions affecting the temporomandibular joint or the masticatory muscles as well as their associated structures. TMD has a prevalence of approximately 10-20% and is 1.5 to 2 times more prevalent in women. It is often associated with restricted mouth opening capacity, pain upon chewing, muscle soreness and headache, thus affecting quality of life considerably although it is not life threatening. The prevalence of reported chronic pain in children and adolescents is high, and similar to the prevalence in adults. The worldwide variation in the prevalence of TMD in children and adolescents ranges from 6% to 69%. Many studies reported that TMD, headache and abdominal pain are the most common chronic pain affecting children and adolescents.

Children and adolescents are treated with routine treatment approaches for adults and one of the most commonly used treatments are occlusal appliances. The use of occlusal appliances in managing orofacial pain conditions is supported by evidence, but only for adults. However, the efficacy of the treatment approaches and any possible side-effects/impairment of mandibular growth are absent. To our knowledge the only two high-quality studies present have investigated adolescents with permanent dentition (12-19 years), but there are no studies in the growing child with primary or mixed dentition (7-14 years). Hence, there is no knowledge if there is an effective treatment and if such a treatment with a resilient occlusal appliance impair the mandibular growth in these children.

Taken together there is immense need for research on treatment of children/adolescents with orofacial pain and following their growth in order to be able to provide effective and safe treatment. Also, to investigate the knowledge-base among care-givers, giving the opportunity to improve the content of the education which in turn would lead to better, faster management of these children/adolescents who actually are our future.

Therefore, the aim of this non-inferiority project is to investigate the effectiveness and possible side-effects of different treatment modalities, such as an occlusal appliance, jaw exercises, NSAID for the conditions myalgia orarthralgia in the orofacial region in children with primary or mixed dentition.

The hypotheses are that: 1) there will be no significant differences in treatment outcome between the use of a soft occlusal appliance and standardized jaw exercises in children with myalgia but that the soft occlusal appliance and the standardized jaw exercises are superior to instructions of self-care; 2) the soft occlusal appliance does not affect the mandibular growth nor the dental eruption pattern; 3) there will be no significant differences in treatment outcome between the use of a soft occlusal appliance, or NSAIDs in children with arthralgia, but that the soft occlusal appliance and the NSAIDs are superior to instructions of self-care.

ELIGIBILITY:
Inclusion Criteria:

* age 7-14 years
* a diagnosis of myalgia or arthralgia according to DC/TMD
* self-assessed average TMD pain intensity of ≥ 30 mm on a 100-mm visual analogue scale (VAS) during one week prior to examination.

The patients will remain included with one or several co-diagnoses of:

* disc displacement with or without reduction according to DC/TMD
* degenerative joint disease.

Exclusion Criteria:

* diagnosed systemic muscular or joint diseases (e.g. fibromyalgia, rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis)
* whiplash associated disorder (WAD)
* neuropathic pain or neurological disorders (e.g. myasthenia gravis, orofacial dystonia)
* history of psychiatric disorders, and 5) pain of dental origin.

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Responders to treatment - median weekly pain intensity | 1-6 months
  30% decrease in median weekly pain intensity using a numeric rating scale 0-10 rating the worst pain daily
Responders to treatment - Patients global impression change scale | 1-6 months
  The patients global impression change scale (PGIC) will be used. PGIC is a 7-point scale with the following options: 0 = eliminated, 1 = much improved, 2 = improved, 3 = unchanged, 4 = impaired, 5 = much impaired and 6 = very much impaired

SECONDARY OUTCOMES:
Change in physical functioning using the Graded Chronic Painscale (GCPS) | 1-6 months
  The graded chronic pain scale include 3 questions regarding pain intensity and 3 questions regarding physical functioning.
  The mean of the 3 questions regarding provide us with the characteristic pain intensity while the mean of the physical functgioning questions together with sick leave (from work/school) provide us with information about how pain affects physical functioning.
  Characteristic pain intensity ranges from 0-100 while physical functioning is graded from 0-IV.
  The lower, the better outcome for all subscales.
  GCPS is a stanrd tool in the Diagnostic Criteria for temporomandibular disorders (DC/TMD) and part of Axis II which also the questionnaires for the emotional status in Oiutcome 3 are.
Change in emotional status | 1-6 months
  Changed scores in questionnaires from Axis II in DC/TMD, including stress using the Perceived Stress Scale-4 (PSS-4), anxiety/depression using the Patient Health Questionnaire-4 (PHQ-4) and the psychosocial situation using the Youth Self-report (YSR) Lower scores in these questionnair represent a better outcome The PSS and PHQ-scales are not combained and ranges from 0-4 for each questions. The YSR is based on several subscales, including the DCM-IV.
Daily activities | 1-6 months
  This outcome is based on a daily question of school attendance as well as free-time activities. The question is did you attend at school today or did you stay at home due to your orofacial pain. Question 2. Did you do your free-time activity or did you stay at hom due to your orofacial pain

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Christidis, PhD, Principal Investigator — Karolinska Institutet, Department of Dental Medicine
Locations (1):
- Karolinska Institutet, Department of Dental Medicine, Huddinge, Sweden